CLINICAL TRIAL: NCT02020564
Title: Speed of Processing Training to Improve Cognition in Traumatic Brain Injury and Mild Cognitive Impairment: A Randomized Clinical Trial
Brief Title: Speed of Processing Training to Improve Cognition in Traumatic Brain Injury and Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director, Neuropsychology & Neuroscience; Director, Traumatic Brain Injury Research, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-755-12
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Traumatic Brain Injury; Mild Cognitive Impairment
Keywords: Processing Speed; Cognition; Intervention; Traumatic Brain Injury; Mild Cognitive Impairment
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): Computerized exercised will be administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Interventions: Behavioral: Speed of Processing Training
- Placebo control group (Placebo Comparator): Computerized exercises will be administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Interventions: Behavioral: Placebo Control

INTERVENTIONS:
Behavioral: Speed of Processing Training
  Arms: Treatment Group
Behavioral: Placebo Control
  Arms: Placebo control group

SUMMARY:
The purpose of this research study is to investigate the effectiveness of a technique designed to improve processing speed (i.e. the amount of time it takes to process information) in a Traumatic Brain Injury (TBI) population. The study is designed to study how well this technique can help people with TBI increase their processing speed and their ability to function better in everyday life.

DETAILED DESCRIPTION:
The current proposal is designed to apply this treatment protocol to a large sample of individuals with moderate to severe TBI with documented impairment in PS. The goals of the trial are to (a) test the efficacy of this treatment protocol within a TBI population, (b) evaluate the impact of the treatment on everyday functioning, (c) evaluate the longer-term efficacy of the treatment, and (d) examine the utility of booster sessions in facilitating longer-term treatment effects. Individuals with moderate to severe TBI, with documented impairment in PS, will be randomly assigned to a treatment group or a control group. Both groups will undergo baseline, immediate post-treatment and long-term follow-up assessment consisting of: (1) a standardized neuropsychological battery and (2) an assessment of global functioning examining the impact of the treatment on daily activities. This design will allow us to assess the efficacy of SPT in persons with TBI and evaluate its impact on everyday life.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Traumatic Brain Injury or Mild cognitive impairment
* Fluent in English
* processing speed impairment

Exclusion Criteria:

* prior stroke or neurological disease
* currently taking steroids and/or benzodiazepines
* history of significant pyschiatric illness (for example, bipolar disorder, schizophrenia, or pyschosis) or a current diagnosis of Major Depressive Disorder, Schizophrenia, Epilepsy, Bipolar Disorder
* significant alcohol or drug abuse history

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-12-12 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Symbol-Digit Modalities Test | Baseline (week 1), immediately post-intervention (week 7) and 3 months post-intervention
  Change in scores on standardized neuropsychological tests of Processing Speed using Symbol-Digit Modalities Test

SECONDARY OUTCOMES:
TBI Quality of Life, Depression scale | Baseline (week 1), immediately post-intervention (week 7) and 3 months post-intervention
  Change in scores on self-report of emotional functioning, measured via questionnaire. The TBI QOL Depression scale measures depression. The range is 1-40. A higher score indicates greater depression.
Perceived Deficits Questionnaire | Baseline (week 1), immediately post-intervention (week 7) and 3 months post-intervention
  Change in scores on self-report of perceived cognitive deficits in daily life, measured via questionnaire. A higher score indicates greater perceived deficits in daily life. Range of scores on the scale is 0-80.
TBI Quality of Life, Total Score | Baseline (week 1), immediately post-intervention (week 7) and 3 months post-intervention
  Change in scores on self-report of quality of life, measured via questionnaire. DV is the TBI-QOL total score. The range is 1-40. A higher score indicates better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Goverover Y, Costa SL, DeLuca J, Chiaravalloti N. Does speed of processing training improve everyday life functional activity in traumatic brain injury: A pilot randomized controlled trial. Neuropsychol Rehabil. 2025 Jul 4:1-16. doi: 10.1080/09602011.2025.2526663. Online ahead of print. PMID 40615123